CLINICAL TRIAL: NCT00348361
Title: A Study to Validate Key Therapeutic Targets and Biomarkers During Allergen Exposure in Subjects With Allergic Rhinitis
Brief Title: Exploration Of Key Targets And Biomarkers Involved In An Allergic Response In Subjects With Allergic Rhinitis (Hay Fever)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Study Director, GSK
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: ELR100710
Record Dates: First submitted 2006-06-30; First posted 2006-07-04 (Estimated); Last update posted 2008-10-13 (Estimated); Status verified 2008-10

CONDITIONS: Allergic Rhinitis
Keywords: Hay fever; biomarkers
MeSH Terms: conditions — Rhinitis, Allergic; Rhinitis, Allergic, Seasonal | interventions — Fluticasone

INTERVENTIONS:
Drug: Fluticasone Propionate

SUMMARY:
This study is aimed at validating key therapeutic targets and biomarkers associated with allergic rhinitis. The therapeutic target expression will be investigated after a 7 day course of corticosteroid treatment followed by allergen challenge.

ELIGIBILITY:
Inclusion criteria:

* No signs or symptoms of rhinitis outside of the relevant airborne allergen season.

Exclusion criteria:

* History or current evidence of an upper or lower respiratory infection or symptoms (including common cold) within 2 weeks of baseline assessments.
* Symptoms of rhinitis at inclusion indicated by total VAS score of >40 for the combined symptoms scores for blockage, rhinorrhoea, sneezing, itching) or a single symptom with a VAS score >20.
* Subjects not showing a nasal response to allergen concentration =< 10,000 BU/ml.
* Subjects with positive skin prick test for Dust House Mite.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48
Dates: Start 2005-04

PRIMARY OUTCOMES:
Change in expression of key allergy targets in the nose following exposure to allergen. Assessment of protein expression measured by western blotting and immunohistochemistry in nasal biopsy tissue.

SECONDARY OUTCOMES:
Effect of corticosteroids treatment on the change in target expression following allergen challenge. Nasal lavage fluid and nasal secretions will be measured by ELISA and chemiluminescent assay.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, MD,MSc, FPPM, Study Director — GlaxoSmithKline
Locations (2):
- GSK Investigational Site, Amsterdam, Netherlands
- GSK Investigational Site, London, London, United Kingdom